CLINICAL TRIAL: NCT02369211
Title: Pharmacoeconomics and Related Patient Outcomes of Multi-dose Intravenous Acetaminophen (OFIRMEV) in Patients Undergoing Robotic-assisted Laparoscopic Prostatectomy
Brief Title: Pharmacoeconomics and Related Patient Outcomes of Multi-dose Intravenous Acetaminophen (OFIRMEV)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Principal Investigator, Richard D Urman, Assistant Professor of Anesthesia, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014P002749
Record Dates: First submitted 2015-02-17; First posted 2015-02-23 (Estimated); Results first posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Prostatectomy; Pain
Keywords: acetaminophen
MeSH Terms: conditions — Pain | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous acetaminophen (Experimental): Patient receives 1g intravenous acetaminophen after the incision
  Interventions: Drug: Acetaminophen (Ofirmev)
- Placebo (Placebo Comparator): Patient receives saline injection instead of the study drug
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Acetaminophen (Ofirmev) — The patient was administered IV Ofirmev during anesthesia and then 3 more IV doses (1g each) every 6 hours up to 24 hrs.
  Other Names: Ofirmev
  Arms: Intravenous acetaminophen
Other: Placebo — The patient was administered IV Placebo during anesthesia and then 3 more doses of IV Placebo every 6 hours up to 24 hrs.
  Arms: Placebo

SUMMARY:
To examine pharmacoeconomics of IV acetaminophen (Ofirmev). Specifically, to examine its potential to improve hospital efficiency and patient outcomes. The investigators compare the addition of IV acetaminophen versus placebo on postoperative anesthesia care unit recovery times, inpatient hospital length of stay (LOS), postoperative pain scores, consumption of opiates as rescue agents and side effects among patients undergoing robotic-assisted laparoscopic prostatectomy (RALP).

DETAILED DESCRIPTION:
Although IV acetaminophen has been studied in urologic surgery, it has not been studied specifically in prostatectomies, and therefore there are no outcomes or cost-effectiveness data currently available. In addition, the current trend is to perform prostatectomy with a robot-assisted laparoscopic technique to help minimize incision size, blood loss, postoperative pain, and speed up patient recovery. Current literature only includes the use of opioids in the perioperative setting for robot-assisted prostatectomy to treat pain, but only a small trial used oral acetaminophen as a measure for analgesia in RALP. In addition to the decreasing use of opioids in perioperative pain management, emphasis has been placed on reducing costs of healthcare. A major contributor to this issue is hospital length of stay (LOS) and there has been increased pressure on healthcare providers to decrease overall LOS. Several factors may contribute to hospital LOS, including hospital acquired infections, surgical recovery, wound care, other surgical and anesthesia-related complications, and importantly, inadequate pain control.

In this study we examine the impact of adding IV acetaminophen to the multimodal analgesic regimen for robotic-assisted laparoscopic prostatectomy (RALP). Our hypothesis is that the addition of IV acetaminophen can improve postoperative recovery time, inpatient LOS, postoperative pain scores, and opioid consumption.

This study specifically addresses pharmacoeconomics of IV acetaminophen. The goal is to understand its potential to improve hospital efficiency and patient outcomes. The study compares the impact of the addition of IV acetaminophen versus a placebo on postoperative anesthesia care unit recovery times, inpatient LOS, postoperative pain scores, consumption of opiates as rescue agents and side effects in patients undergoing RALP.

The study is a 2-arm, double-blind, randomized, placebo controlled trial comparing IV acetaminophen to a control (IV placebo). All patients in this study were scheduled to undergo RALP.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing robotic-assisted laparoscopic prostatectomy
* ≥18 years old males
* American Society of Anesthesiologists class 1-4

Exclusion Criteria:

* Chronic opiate use
* Liver disease (known history of hepatitis B or C, cirrhosis, nonalcoholic steatohepatitis, history of alcoholism, liver function test results greater than 3 times upper limit of normal in the past 3 months)
* Allergy/hypersensitivity to acetaminophen
* Patients with baseline dementia
* Chronic diathesis
* Chronic kidney disease

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Urman, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in the preoperative assessment clinic prior to undergoing surgery
Groups:
- Intravenous Acetaminophen: Patient receives 1g intravenous acetaminophen after the incision
  Acetaminophen (Ofirmev)
- Placebo: Patient receives saline injection instead of the study drug
  Placebo
Period: Overall Study
Arm/Group | Intravenous Acetaminophen | Placebo
Started | 43 | 43
Completed | 43 | 41
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Population: analysis population is the same as the assignment in Participant flow
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Acetaminophen | Placebo | Total
Number analyzed (Participants) | 43 | 41 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 16 | 30
  >=65 years | 29 | 25 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (6.1) | 60.2 (6.3) | 61.7 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 43 | 41 | 84
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 43 | 41 | 84

OUTCOME MEASURES:

1. Primary Outcome: Post Anesthesia Care Unit Length of Stay
Description: The amount of time patients stayed in the post-anesthesia care unit following anesthesia, before going to the inpatient ward.
Time Frame: approximately 30-240 min
Population: Patients who had surgery and were then transferred to the post-anesthesia care unit for recovery.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Intravenous Acetaminophen | Placebo
Number analyzed (Participants) | 34 | 41
minutes | 124 (58.26) | 132 (62.58)

2. Primary Outcome: Hospital Length of Stay
Description: This outcome measure calculates the number of days the patient stayed in the hospital before being discharged home.
Time Frame: 1-3 days
Population: Patients who were admitted to the hospital (as inpatients) following surgery and post-anesthesia care unit stay.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Intravenous Acetaminophen | Placebo
Number analyzed (Participants) | 34 | 41
Days | 0.81 [0.71 to 0.90] | 0.82 [0.66 to 0.95]

3. Secondary Outcome: Pain Score
Description: Pain scores were collected using the Visual Analog Scale. The scale range is 0 (no pain) to 10 (most pain).
  Mean pain score over first 24 hours postoperatively was collected.
Time Frame: 0-24 hours after surgery
Population: Patients who were assessed for levels of pain following surgery, including both treatment and placebo arms.
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intravenous Acetaminophen | Placebo
Number analyzed (Participants) | 41 | 43
score on a scale | 0.62 [0.13 to 1.00] | 0.88 [0.38 to 2.00]

4. Secondary Outcome: Opioid Use
Description: A measure of the amount of opioid study patients used postoperatively while recovering from surgery at the hospital
Time Frame: 0-24 hours
Population: Patients who underwent surgery and stayed in the hospital as inpatients and received pain management.
Measure: Median (Inter-Quartile Range); unit: morphine milligram equivalents
Arm/Group | Intravenous Acetaminophen | Placebo
Number analyzed (Participants) | 43 | 41
morphine milligram equivalents | 42 [36.4 to 50.0] | 50 [35.6 to 72.0]

ADVERSE EVENTS:
Time Frame: Patients were followed for 30 days after surgery for which adverse events were collected.
Description: Same definition of adverse event was used.
Arm/Group | Intravenous Acetaminophen | Placebo
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/41
Other Adverse Events (participants affected / at risk) | 0/43 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-16): https://cdn.clinicaltrials.gov/large-docs/11/NCT02369211/Prot_SAP_000.pdf